CLINICAL TRIAL: NCT06872723
Title: CPRIT: Patient Adherence to Lung Cancer Screening
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1489
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung Cancer Screening: Participants who agree to take part in this study, will participate in an interview. During the interview, participants may be asked about:
  * Participants background information, such as your race and level of education
  * Participants lung cancer diagnosis and your history of lung cancer screening
  * Participants experience with scheduling lung cancer screening
  * Any barriers that kept participants from completing screening
  Interventions: Behavioral: Lung Cancer Screening

INTERVENTIONS:
Behavioral: Lung Cancer Screening — Participants who agree to take part in this study, will participate in an interview. During the interview, participants may be asked about: • Participants background information, such as your race and level of education • Participants lung cancer diagnosis and your history of lung cancer screening • Participants experience with scheduling lung cancer screening • Any barriers that kept participants from completing screening

SUMMARY:
To understand participants' barriers to lung cancer screening and their experience with scheduling lung cancer screening.

DETAILED DESCRIPTION:
Primary Objectives/Aims

1. Determine rates of lung cancer scheduling and screening at the UTMB and UT Tyler LCS programs.
2. Using state-of-the-art machine learning (ML) approaches, develop prediction models for adherence to screening guidelines for newly eligible and established patients. Investigators will leverage data from BRFSS, UT Tyler and UTMB to develop and validate the prediction model, ensuring its generalizability and accuracy.
3. Survey participants in the LCS programs about their impressions and experience with the scheduling and completing screening; conduct interviews with participants who receive an order for LCS but do not complete screening by their due date.
4. Interview LCS program directors and staff about barriers and facilitators of increasing screening rates in their programs.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker or quit within the past 15 years
* A 20+ pack-year smoking history
* Healthy enough for treatment

Exclusion Criteria:

* Not applicable as our focus is on patients with an order for screening at the UTMB or UT Tyler

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Volk, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT06872723/ICF_000.pdf